CLINICAL TRIAL: NCT00671658
Title: Phase II Study of The Modified Hyper-CVAD Program for Acute Lymphoblastic Leukemia
Brief Title: Modified Hyper-CVAD (Cyclophosphamide, Vincristine, Adriamycin, and Dexamethasone) Program for Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID02-230
Record Dates: First submitted 2008-04-30; First posted 2008-05-05 (Estimated); Results first posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Leukemia; Acute Lymphoblastic Leukemia
Keywords: Lymphoma; HYPER-CVAD; Leukemia; Acute Lymphoblastic Leukemia; ALL; Remission Duration; Chemotherapy; Asparaginase; Cyclophosphamide; Cytarabine; Dexamethasone; Doxorubicin; Leukine; Methotrexate; Rituximab; Vincristine
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Dexamethasone; Calcium Dobesilate; Methotrexate; Cytarabine; Granulocyte Colony-Stimulating Factor; Filgrastim; Mesna; pegaspargase; pegfilgrastim; pegylated granulocyte colony-stimulating factor, human; Methylprednisolone Hemisuccinate; Methylprednisolone; Methylprednisolone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HYPER-CVAD (Experimental): Rituximab 375 mg/m^2 intravenous (IV), Cyclophosphamide (CTX) 300 mg/m^2 IV, Doxorubicin 50 mg/m^2 IV, Vincristine 2 mg IV, Dexamethasone 40 mg IV or oral (PO). Methotrexate (MTX) 12 mg intrathecally (6 mg if via Ommaya reservoir) for Courses 1,3,5,7 - 200 mg/m^2 IV followed by 800 mg/m^2 for Courses 2,4,6,8. Cytarabine 100 mg intrathecal for Courses 1,3,5,7 - 3 gm/m^2 IV for Courses 2,4,6,8. G-CSF 10 ug/kg subcutaneous injection. Mesna 600 mg/m2 a day IV, Pegylated asparaginase 2000 International units/m^2 IV. Pegfilgrastim 6 mg (flat dose) within 72 hrs after completion of chemotherapy. Solumedrol 40 mg IV for Courses 2,4,6,8.
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide (CTX); Drug: Doxorubicin; Drug: Vincristine; Drug: Dexamethasone; Drug: Methotrexate (MTX); Drug: Cytarabine; Drug: G-CSF; Drug: Mesna; Drug: Pegylated asparaginase; Drug: Pegfilgrastim; Drug: Solumedrol

INTERVENTIONS:
Drug: Rituximab — 375 mg/m2 by vein
  Other Names: Rituxan
Drug: Cyclophosphamide (CTX) — 300 mg/m2 by vein
  Other Names: Cytoxan; Neosar
Drug: Doxorubicin — 50 mg/m2 by vein
  Other Names: Adriamycin; Rubex
Drug: Vincristine — 2 mg by vein
  Other Names: Oncovin; Vincasar Pfs
Drug: Dexamethasone — 40 mg by vein or by mouth (P.O.)
  Other Names: Decadron
Drug: Methotrexate (MTX) — 12 mg intrathecally (6 mg if via Ommaya reservoir) for Courses 1,3,5,7
  200 mg/m2 by vein followed by 800 mg/m2 for Courses 2,4,6,8
  Other Names: Rheumatrex
Drug: Cytarabine — 100 mg intrathecal for Courses 1,3,5,7
  3 gm/m2 by vein for Courses 2,4,6,8
  Other Names: Ara-C; Cytosar-U; Arabinosylcytosine; DepoCyt
Drug: G-CSF — 10 ug/kg subcutaneous injection
  Other Names: Filgrastim; Neupogen
Drug: Mesna — 600 mg/m2 a day by vein
  Other Names: Mesnex
Drug: Pegylated asparaginase — 2000 International units/m2 by vein
  Other Names: Pegaspargase; Oncaspar; Polyethylene Glycol Conjucated Lasparaginase-H
Drug: Pegfilgrastim — 6 mg (flat dose) within 72 hrs after completion of chemotherapy
  Other Names: Neulasta; PEG-G-CSF
Drug: Solumedrol — 40 mg by vein for Courses 2,4,6,8
  Other Names: Methylprednisolone; Depo-Medrol; Medrol

SUMMARY:
The goal of this clinical research study is to learn if intensive chemotherapy (with monoclonal antibody therapy in some patients) given for 8 courses over 5 to 6 months followed by monthly maintenance chemotherapy for 2 ½ years can improve or cure acute lymphoblastic leukemia (ALL) or lymphoblastic lymphoma.

DETAILED DESCRIPTION:
The modified hyper-CVAD regimen is a combination of chemotherapy drugs including cyclophosphamide, vincristine, Adriamycin, dexamethasone and pegylated asparaginase given together for one "course" of treatment. This alternates with a course or combination of the chemotherapy drugs methotrexate, cytarabine (ara-C), and pegylated asparaginase. Rituximab is a protein (monoclonal antibody) that attaches to the surface of the leukemia or lymphoma cells, which have a marker, called "CD20".

Before treatment starts, participants will have a complete physical exam, including blood (about 8 teaspoons) tests. A chest X-ray may be taken. CT scans may be taken if needed. A bone marrow sample will be taken through a large needle in the hipbone. Women able to have children must have a negative blood pregnancy test. An ECG (tracing of the heart) and a cardiac scan or echocardiogram may be taken to check the heart function.

Participants will receive these 2 kinds of intensive chemotherapy courses for a total of 8 courses as long as they are able to tolerate them. Chemotherapy courses will be given through a large vein by a central venous catheter (a plastic tube usually placed under the collarbone) or a long-line catheter (a plastic tube usually placed in the upper arm).

During treatment, participants will have a physical exam and undergo blood tests (about 1 tablespoon each) at least twice a week. After the first course of chemotherapy, the tests done before treatment will be repeated to check for response. In patients with acute lymphoblastic leukemia or lymphoblastic lymphoma with marrow disease, a bone marrow sample will be repeated about 2 and 3 weeks from the beginning of treatment to check the response.

Course 1 (odd courses) will start by giving rituximab by vein over 6 hours on Day 1 and Day 11 for patients whose leukemia or lymphoma expresses CD20. Participants will receive the drugs acetaminophen (Tylenol) and diphenhydramine hydrochloride (Benadryl) 30-60 minutes before each dose of rituximab. This will be done to lessen the risk of fever, chills, and allergic reactions. Usually, the first dose of rituximab requires about 6 to 8 hours to complete. If side effects do occur during the infusion, participants will be observed for an additional 2 hours after the rituximab is given. Then, the cyclophosphamide will be given as described below.

Other participants who do not have the CD20 marker will start Course 1 with cyclophosphamide given by vein over 2-3 hours every 12 hours. This will be given for 6 doses over 3 days (Days 1,2, and 3). Pegylated asparaginase will be given by vein over 30 minutes on Day 1. Adriamycin will be given by vein over 24 hours on Day 4. Vincristine will be given by vein over 15 to 30 minutes on Days 1 and 11. Dexamethasone (a steroid) will be given by mouth or by vein on Days 1 to 4 and 11 to 14.

Pegfilgrastim (a growth colony stimulating factor) will be given after each course of chemotherapy is finished. It is given to help with rapid recovery of the white blood cells in the normal marrow. Pegfilgrastim will be injected under the skin within 72 hours of completion of each cycle of chemotherapy. Filgrastim, a shorter active form of pegfilgrastim may be used instead or added later if needed.

Treatment to protect the brain will be given inside the spinal using lumbar punctures (spinal taps) with chemotherapy, including methotrexate around day 2 and cytarabine (ara-C) about day 7 of the course. This is done to decrease the risk that the leukemia or lymphoma will develop there. If there is leukemia or lymphoma in the spinal fluid at the time of the first spinal tap, then the treatments will be given more frequently.

For patients aged 60 years or older, this first course of chemotherapy will be given in a protective isolation room to decrease the risk of infection(s).

During Course 2, participants whose leukemia expresses CD20 will receive rituximab by infusion over 4 hours on Days 1 and 8. Other participants who do not have CD20 on the leukemia cells will start with methotrexate by vein over 24 hours on Day 1. Cytarabine (ara-C) will be given by vein over 2 hours every 12 hours for 4 doses (Days 2 and 3). Vincristine will be given by vein over 15 to 30 minutes on Days 1 and 8. Pegylated asparaginase will be given by vein over 30 minutes on Day 4 or 5 after the methotrexate has cleared (as checked by blood tests).

Citrovorum factor (leucovorin), an antidote for side effects of methotrexate, will be given by vein or by mouth for 2-3 days (Day 2 and on). Pegfilgrastim will be given as in Course 1 (24-72 hours after the chemotherapy is finished). The treatment to protect the brain inside the spinal fluid will be given as in Course 1 on Days 2 and 7.

The rest of the chemotherapy will switch between hyper-CVAD and pegylated asparaginase (Courses 3, 5, and 7) and methotrexate,cytarabine (ara-C), vincristine, and pegylated asparaginase (Courses 4, 6, and 8) to complete a total of 8 courses. Participants whose leukemia expresses CD20 will receive a total of 12 doses (2 per each of the first four courses, then one with the last four courses) of rituximab.

After the 8 courses, patients with lymphoblastic lymphoma who had enlarged lymph glands in the mediastinum may receive radiation to the chest. Those participants not needing radiation will proceed to monthly maintenance chemotherapy. This includes daily 6-mercaptopurine taken by mouth, weekly methotrexate by vein or mouth, monthly vincristine by vein, and dexamethasone by mouth for 5 days every month. Participants with lymphoblastic lymphoma will start maintenance chemotherapy after finishing radiation.

Maintenance chemotherapy will be given for a total of 30 months, and will be interrupted by 2 periods of intensive chemotherapy courses. The first will be at six months into the maintenance program starting first with hyper-CVAD (like Course 1) except without pegylated asparaginase). The following months, participants will receive methotrexate by vein on Day 1, vincristine by vein on Day 1, and pegylated asparaginase by vein on Day 2. Participants will receive this sequence of 2 chemotherapy courses again 18 months into the maintenance program. Participants with the CD20 marker will receive rituximab during the maintenance chemotherapy (with the vincristine during months 1, 3, 6, 7, 10, 13, 18 & 19).

After one or two courses of therapy, the response to the treatment will be evaluated. If the leukemia or lymphoma is responding, the therapy will be continued. Participants will be taken off study if the leukemia or lymphoma starts to get worse.

After completion of treatment, participants will have a complete physical exam, including blood tests (about 8 teaspoons). If needed, a chest X-ray or CT scan will be done. A bone marrow sample will be taken through a large needle. Patients will then return every 3 to 6 months for a checkup, including blood tests and bone marrow aspiration. X-rays may be repeated if needed.

An Ommaya reservoir may also be placed surgically as a route to treat leukemia in the brain or to decrease the risk of leukemia in patients who have difficulty with the spinal treatments. An Ommaya reservoir is a tube inserted under the skin of the scalp that enters into the spinal fluid cavity of the brain.

Treatment will be given on an inpatient basis for the 8 intensive cycles of chemotherapy, or as indicated by the clinical condition. The maintenance treatments will be given as an outpatient but may be given as an inpatient if needed.

This is an investigational study. All of the drugs are commercially available. Their use together in this study is investigational. About 280 patients will take part in this study. All will be enrolled at M. D. Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed, previously untreated Acute Lymphoblastic Leukemia (ALL) or lymphoblastic lymphoma, or having achieved Complete Remission (CR) with one course of induction chemotherapy.
2. Failure to one induction course of chemotherapy are eligible, but these patients will be analyzed separately.
3. All ages are eligible.
4. Zubrod performance less than or equal to 3
5. Adequate liver function (bilirubin </= 3.0 mg/dl unless considered due to tumor) and renal function (creatinine </= 3.0 mg/dl, unless considered due to tumor).
6. Adequate cardiac function as assessed by history and physical examination.
7. No active co-existing malignancy with life expectancy less than 12 months due to that malignancy.

Exclusion Criteria:

1) N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2002-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan O'Brien, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Official Website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 11/02/2002 to 8/28/2012. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Groups:
- HYPER-CVAD: Rituximab 375 mg/m^2 intravenous (IV), Cyclophosphamide (CTX) 300 mg/m^2 IV, Doxorubicin 50 mg/m^2 IV, Vincristine 2 mg IV, Dexamethasone 40 mg IV or oral (PO). Methotrexate (MTX) 12 mg intrathecally (6 mg if via Ommaya reservoir) for Courses 1,3,5,7 - 200 mg/m^2 IV followed by 800 mg/m^2 for Courses 2,4,6,8. Cytarabine 100 mg intrathecal for Courses 1,3,5,7 - 3 gm/m^2 IV for Courses 2,4,6,8. G-CSF 10 ug/kg subcutaneous injection. Mesna 600 mg/m^2 a day IV, Pegylated asparaginase 2000 International units/m^2 IV. Pegfilgrastim 6 mg (flat dose) within 72 hours after completion of chemotherapy. Solumedrol 40 mg IV for Courses 2,4,6,8.
Period: Overall Study
Arm/Group | HYPER-CVAD
Started | 220
Completed | 215
Not Completed | 5
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Arm/Group | HYPER-CVAD
Number analyzed (Participants) | 220
Age, Continuous [Median (Full Range); unit: years] | 46 [16 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102
  Male | 118
Region of Enrollment [Number; unit: participants]
  United States | 220

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Response
Description: Response - Complete remission (CR): Normalization peripheral blood & bone marrow 5% or <blasts in normocellular or hypercellular marrow granulocyte count of 1x10^9/L or > & platelet count >100x10^9/L; CR with incomplete platelet recovery (CRp): CR but platelet count <100x10^9/L. CR with incomplete recovery (CRi): CR but platelet count <100x10^9/L or absolute neutrophil count < 1x10^9/L. Partial response (PR): As above except for presence of 6-25% marrow blasts. Lymphoblastic lymphoma (& ALL subtypes with extramedullary disease): CR - disappearance all known disease. PR - >50% decrease in tumor size using sum of product, includes 50% volume decrease in lesions measurable in 3 dimensions. No Response (NR) - No significant change (includes stable disease). Lesions decreased size but <50% or lesions with slight enlargement <25% increase in size. Progressive Disease (PD): Appearance new lesions, 25% or > increase in size existing lesions (>50% if 1 lesion & <2).
Time Frame: Response assessed following first 21 day course up to end of treatment with 8 cycles, up to 210 days
Measure: Number; unit: Participants
Arm/Group | HYPER-CVAD
Number analyzed (Participants) | 215
Participants
  Complete Response (CR) | 198
  Complete Response without Platelet Recovery | 3
  Partial Response (PR) | 4

ADVERSE EVENTS:
Time Frame: Up to 8 cycles of 21 days with 7 day waiting period in between (approximately 28 days) then 30 following last treatment, therefore up to 210 days for completed treatment periods.
Arm/Group | HYPER-CVAD
All-Cause Mortality (participants affected / at risk) | 25/215
Serious Adverse Events (participants affected / at risk) | 61/215
Other Adverse Events (participants affected / at risk) | 24/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HYPER-CVAD (N=215)
Vision Loss (Eye disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Neutropenic Fever (Infections and infestations) | 34 (60)
Hemorrhage CNS (Blood and lymphatic system disorders) | 1 (1)
Nausea/Vomiting (Gastrointestinal disorders) | 3 (3)
Infection (Infections and infestations) | 32 (54)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Memory Impairment (Nervous system disorders) | 1 (1)
Psychosis (Nervous system disorders) | 1 (1)
Seizures (Nervous system disorders) | 2 (2)
Paraparesis (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypotension (Cardiac disorders) | 3 (3)
Pain (General disorders) | 7 (7)
Syncope (Nervous system disorders) | 4 (5)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Blurred Vision (Eye disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Acute Pancreatitis (Hepatobiliary disorders) | 2 (2)
Arm Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Death (General disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hydro-Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Soft Tissue Necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Fibrinogen decreased (Blood and lymphatic system disorders) | 1 (1)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Flu-Like Syndrome (General disorders) | 2 (2)
Neuropathy (Nervous system disorders) | 2 (2)
Thrombosis Embolism (Vascular disorders) | 1 (1)
Abdominal Pain (General disorders) | 4 (4)
Acute Cholecystitis (Hepatobiliary disorders) | 1 (1)
Acute Renal Failure (Renal and urinary disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Back Pain (General disorders) | 3 (3)
Bactremia (Blood and lymphatic system disorders) | 1 (2)
Bronchitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Chest Pain (General disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Duodenal Ulcer (Gastrointestinal disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 2 (2)
Fever (General disorders) | 4 (5)
Gastrointestinal Rectum Hemorrhage (Gastrointestinal disorders) | 1 (1)
Hemorrhage Gastrointestinal (Gastrointestinal disorders) | 1 (2)
Kidney Stones (Renal and urinary disorders) | 1 (1)
Lung Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Musculoskeletal Soft tissue discomfort (Skin and subcutaneous tissue disorders) | 1 (1)
Pain Gallbladder (General disorders) | 3 (3)
Partial Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1)
Perforated Sigmoid Colon (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Renal Failure (Renal and urinary disorders) | 1 (1)
Right Eye Retinal Necrosis (Eye disorders) | 1 (1)
Right Subclavian Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HYPER-CVAD (N=220)
Diarrhea (Gastrointestinal disorders) | 10 (10)
Neutropenic Fever (Infections and infestations) | 24 (24)
Infection (Infections and infestations) | 20 (20)
Neutropenia (Blood and lymphatic system disorders) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes